CLINICAL TRIAL: NCT00792857
Title: Single-Dose, Two-Period, Open Label, Dose Determination, Randomized, Cross-Over Study of CTAP201 Injection and Doxercalciferol (Hectorol) Injection in Subjects With Stage 5 CKD and SHPT on Hemodialysis
Brief Title: Comparison of I.V. CTAP201 and Doxercalciferol (Hectorol) in Subjects With Chronic Kidney Disease (CKD) and Secondary Hyperparathyroidism (SHPT)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO IP Holdings II, Inc. (Industry)
Responsible Party: Sponsor
Organization: OPKO Health, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTAP201-CL-1007
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Kidney Disease; Secondary Hyperparathyroidism; Chronic Renal Insufficiency; Chronic Renal Failure
Keywords: Parathyroid Diseases; Renal Insufficiency; Kidney Failure, Chronic; Hyperparathyroidism, Secondary; Vitamin D; Hyperparathyroidism; Renal Insufficiency, Chronic; Kidney Diseases; Kidney Failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary; Kidney Failure, Chronic; Parathyroid Diseases; Renal Insufficiency; Hyperparathyroidism; Kidney Diseases | interventions — 1 alpha-hydroxyergocalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CTAP201 Injection at dose a (Experimental): CTAP201 at dose a
  Interventions: Drug: CTAP201 Injection
- CTAP201 Injection (Experimental): CTAP201 at dose b or dose c
  Interventions: Drug: CTAP201 Injection
- Doxercalciferol at dose a (Active Comparator): Active at dose a
  Interventions: Drug: Doxercalciferol
- Doxercalciferol (Active Comparator): Active at dose b or dose c
  Interventions: Drug: Doxercalciferol

INTERVENTIONS:
Drug: CTAP201 Injection — Comparison of different dose strengths of CTAP201 after single dose.
  Arms: CTAP201 Injection; CTAP201 Injection at dose a
Drug: Doxercalciferol — Comparison of different dose strengths of doxercalciferol after single dose.
  Other Names: Hectorol
  Arms: Doxercalciferol; Doxercalciferol at dose a

SUMMARY:
This study will compare CTAP201 with Doxercalciferol in patients with chronic kidney disease (CKD) and secondary hyperparathyroidism (SHPT), undergoing regular hemodialysis, at different dose strengths. This study will also investigate the levels of CTAP201 in the body over time and determine the safety of CTAP201.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 40
* On maintenance hemodialysis three times per week
* Visit 1: Serum iPTH value greater than or equal to 200 pg/mL and lower than or equal to 1000 pg/mL
* Visit 1: Serum total calcium value greater than 8.4 mg/dL and lower than 10.0 mg/dL
* Visit 1: Serum phosphorus value greater than or equal to 2.5 mg/dL and lower than or equal to 5.5 mg/dL
* Serum 25-hydroxyvitamin D level greater than or equal to 15 ng/mL
* Visit 2: Serum iPTH value greater than 300 pg/mL
* Visit 2: Serum Ca x P product less than 56 [mg/dl]2
* Willing and able to discontinue vitamin D and/or bone metabolism therapy for at least 2 weeks prior to administration of Study Drug, and length of study

Exclusion Criteria:

* Taking cytochrome P450 3A inhibitors and/or inducers
* Abnormal liver functions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Blood levels of CTAP201 and doxercalciferol | Day 1 and Day 15 of each dose level
Safety of a single dose of CTAP201 Injection | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Joel Melnick, MD, Study Director — OPKO Renal
Locations (6):
- United States (6):
  - Pivotal Reseach Centers, Peoria, Arizona
  - Western New England Renal and Transplant Associates, Springfield, Massachusetts
  - University of Cincinnati, Cincinnati, Ohio
  - Northeast Clinical Research, Allentown, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Southwest Houston Research Ltd., Houston, Texas